CLINICAL TRIAL: NCT06321055
Title: Real-World Regorafenib Use Among Advanced Gastrointestinal Stromal Tumors
Brief Title: An Observational Study to Learn More About Treatment With Regorafenib in People With Advanced Gastrointestinal Stromal Tumors in the United States
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22533
Record Dates: First submitted 2024-03-14; First posted 2024-03-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Advanced Gastrointestinal Stromal Tumor
MeSH Terms: interventions — regorafenib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Advanced Gastro-intestinal soft-tissue tumors (GIST) patients: Adult GIST patients with evidence of regorafenib treatment initiation among commercially insured or Medicare patients in the Merative MarketScan database.
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — Retrospective analysis.

SUMMARY:
This is an observational study in which data already collected from people with advanced gastrointestinal stromal tumors are studied.

In this observational study data are collected from participants who have private insurance or Medicare and who had started regorafenib treatment.

Gastrointestinal stromal tumor (GIST) is a type of cancer that most commonly originates from the stomach or small intestine. Advanced means that the cancer has spread to other parts of the body.

The study drug, regorafenib, is already approved for doctors to prescribe to people with GIST. Regorafenib works by blocking certain proteins that cause the growth of cancer cells. Regorafenib is recommended as the third choice of treatment for patients after imatinib and sunitinib have stopped working or have caused side effects that are too severe to continue the treatment. In addition, it is also the recommended first choice of treatment in people with GIST who had low levels of protein called succinate dehydrogenase (SDH) protein. This condition is called SDHdeficient GIST. However, doctors might sometimes give it in a different order. To better understand the treatment patterns with regorafenib for GIST, more knowledge is needed about its use in the real world.

The participants in this study had started treatment with regorafenib as part of their regular care from their doctors.

The main purpose of this study is to learn more about the use of regorafenib treatment among people with advanced GIST who have private insurance or Medicare in the United States. To do this, researchers will collect information on:

Duration of treatment with regorafenib (also known as duration of therapy)

The length of time it took for participants to switch to another GIST treatment after starting regorafenib (also known as time to next therapy)

The data will come from the participants' information stored in a database, called Merative MarketScan for people in the United States. Data collected will be from April 2002 to September 2023.

Researchers will track the data of people with GIST who started regorafenib and will follow them for at least 28 days.

In this study, only available data are collected. No visits or tests are required as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if they:

  1. Have evidence of ≥1 pharmacy claim for regorafenib during the identification period from 1 October 2015, through 30 November 2022 The first prescription claim date for regorafenib during the identification period will be designated as the index date
  2. Have evidence of ≥1 medical claim with GIST diagnosis codes defined by International Classification of Diseases, 10th Revision, Clinical Modification (ICD-10-CM) diagnosis codes any time during the baseline period (establish a GIST diagnosis prior to regorafenib initiation- primary analysis)
  3. Have evidence of ≥1 medical claim with GIST diagnosis codes defined by International Classification of Diseases, 10th Revision, Clinical Modification (ICD-10-CM) diagnosis codes any time during the patient identification period (capture all regorafenib patients with GIST diagnosis in the database- sensitivity analysis)
  4. Have ≥12 months of continuous health plan enrollment prior to the index date, not including the index date
  5. Have ≥28 days of continuous health plan enrollment after the index date, including the index date

     Exclusion Criteria:
* Patients will be excluded if they:

  1. Are aged <18 years as of the index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult GIST patients with evidence of regorafenib treatment initiation among commercially insured or Medicare patients in the Merative MarketScan database.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Duration of Therapy (DOT) on regorafenib | Retrospective analysis from 1 April 2002 to 30 September 2023
Time to Next Therapy (TTNT) therapy after regorafenib | Retrospective analysis from 1 April 2002 to 30 September 2023

SECONDARY OUTCOMES:
Number of the guideline-listed medications other than regorafenib | Retrospective analysis from 1 April 2002 to 30 September 2023
  * Imatinib (Gleevec)
  * Sunitinib (Sutent)
  * Dasatinib (Sprycel)
  * Avapritinib (Ayvakit)
  * Larotrectinib (Vitrakvi)
  * Entrectinib (Rozlytrek)
  * Ripretinib (Qinlock)
  * Dabrafenib (Tafinlar)
  * Trametinib (Mekinist)
  * Cabozantinib (Cabometyx)
  * Nilotinib (Tasigna)
  * Pazopanib (Votrient)
  * Sorafenib (Nexavar)
  * Everolimus in combination with tyrosine kinase inhibitors (Afinitor, Zortress)
  * Ponatinib (Iclusig)
  * Binimetinib (Mektovi)
Descriptive analysis of baseline demographic | Retrospective analysis from 1 April 2002 to 30 September 2023
Descriptive analysis of clinical characteristics | Retrospective analysis from 1 April 2002 to 30 September 2023
Number of patients with evidence of any metastasis on or after the index date during the follow-up period. | Retrospective analysis from 1 April 2002 to 30 September 2023
Number of patients with evidence of surgery on or after the index date during the follow-up period using Current Procedural Terminology (CPT) codes and International Classification of Disease 9/10 Procedure codes (ICD-PC). | Retrospective analysis from 1 April 2002 to 30 September 2023

CONTACTS AND LOCATIONS:
Locations (1):
- Bayer, Whippany, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.